CLINICAL TRIAL: NCT05384821
Title: Phase 1-2 Trial Evaluating Metronomic Chemotherapy in Patients With a Relapsed or Refractory Wilms Tumor
Brief Title: Metronomic Chemotherapy in Wilms Tumor (MetroWilms-1906)
Acronym: MetroWilms
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MetroWilms-1906
Record Dates: First submitted 2021-11-08; First posted 2022-05-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Wilms Tumor
Keywords: Multidrug chemotherapy; metronomic chemotherapy; Wilms Tumor; Renal cancer
MeSH Terms: conditions — Wilms Tumor; Kidney Neoplasms | interventions — Vincristine; Irinotecan; Temozolomide; Etoposide; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm - Vincristine + Irinotécan + Témozolomide + Etoposide + Cis-Retinoic acid (Experimental): Metronomic chemotherapy : Vincristine + Irinotécan + Témozolomide + Etoposide + Cis-Retinoic acid
  Interventions: Drug: Vincristine; Drug: Irinotecan; Drug: Temozolomide; Drug: Etoposide; Drug: Cis-Retinoic acid

INTERVENTIONS:
Drug: Vincristine — IV, D1-D22-D43 and D64
Drug: Irinotecan — Oral, 5 days/week during W1,W2,W7 and W8 (D1 to D5, D8 to D12, D43 to D47, D50 to D54)
Drug: Temozolomide — Oral,3 weeks in a row, twice per cycle (D1 to D21, D43 to D63)
Drug: Etoposide — Oral, 3 weeks in a row, twice per cycle (D22 to D42, D64 to D84)
Drug: Cis-Retinoic acid — Oral, 2 weeks in a row, thrice per cycle (D15 to D28, D43 to D56, D71 to D84)

SUMMARY:
This is a multicenter, interventional, non-randomized study among patients with a relapsed or refractory Wilms tumor. The study will aim to assess efficacy of metronomic chemotherapy, in terms of disease control after two cycles of metronomic chemotherapy.

DETAILED DESCRIPTION:
The main aim of this study is to assess efficacy of metronomic chemotherapy, in terms of disease control after two cycles of metronomic chemotherapy .

Other objectives of the study include:

* To evaluate disease control obtained with metronomic chemotherapy, in terms of progression-free survival (PFS) and overall survival (OS).
* Evaluating early response after one cycle of treatment of metronomic treatment;
* Evaluating best tumor response over the whole metronomic treatment duration;
* Evaluating safety of the proposed metronomic chemotherapy;
* Evaluating the feasibility of the proposed metronomic chemotherapy.
* To evaluate quality of life using Kindl® Quality of Life questionnaire at baseline (before start of treatment), and approximately at weeks 7 and 13 of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 months old and ≤ 17 years old
* Relapsed or refractory Wilms tumor, histologically proven at diagnosis
* After at least 2 lines of chemotherapy (conventional or high dose, which may include the trial molecules) or after 1 line for high risk relapse for which there would not be any curative therapy. If 1 line for high risk relapse, the enrolment should be confirmed by coordinators.
* Radiologically measurable or evaluable disease (visible, target or non-target-lesion on MRI or CT-scan)
* Performance status: Karnofsky performance status (for patients >16 years of age) or Lansky Play score (for patients ≤16 years of age) ≥ 70%.
* Able to take oral medication or nasal gastric tube or authorized gastrostomy
* Adequate biological criteria:

  * Neutrophils > 1000/mm3 ; Platelets > 75 000/mm3
  * Transaminases (ALT/ AST) ≤ 3 times ULN (or ≤ 6 times ULN if liver metastasis); total bilirubin ≤ 2 ULN (except in case of Gilbert's disease)
* Creatinine ≤ 1,5 ULN or clearance ≥ 60 mL/ min/ 1,73m2 (In case of doubt, to be confirm by assessment of cystatin )
* Females of childbearing potential must have a negative seric pregnancy test within 7 days prior to initiation of treatment.
* Sexually active patients must agree to use adequate and appropriate contraception (at least one highly effective contraception or two complementary methods of contraception), 1 month before beginning of treatment while on trial drug and for 7 months after stopping the trial drug for female patients and after 6 months for male patients.
* Written informed consent from parents/legal representative, patient, and age-appropriate assent before any trial-specific screening procedures according to national guidelines.
* Patient covered by the French "Social Security" regime

Exclusion Criteria:

* Prior history of other cancer within 5 years
* Chemotherapy or radiotherapy of target lesion within 3 weeks prior to inclusion
* Target therapy within less than 5 * half-life of the substance prior to inclusion
* Major surgery within 15 days prior to inclusion
* Presence of any NCI-CTCAE v5 grade ≥ 2 cardiac, hepatic, pulmonary or renal toxicity
* Severe myelosuppression
* Severe peripheral neuropathy (grade ≥ 2)
* Fructose intolerance
* Inflammatory bowel chronic disease and/or intestinal obstruction
* Patients with demyelinating form of Charcot-Marie-Tooth disease
* Known active viral hepatitis or known human immunodeficiency virus (HIV) infection or any other uncontrolled infection.
* Known hypersensitivity to dacarbazine (DTIC), isotretinoin or to any of the trial drugs, trial drug classes, excipients in the formulation
* Hyperlipidemia and hypervitaminosis A
* Vaccination with a live attenuated vaccine within 1 month prior to inclusion
* Pregnant or breastfeeding patients
* Inability to comply with medical follow-up of the trial (geographical, social or psychological reasons)

Ages: 18 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Disease control | 6 months after inclusion
  Complete response, partial response or stable disease after 2 cycles of treatment, measured by the progression-free survival (PFS).

SECONDARY OUTCOMES:
Progression-free survival | Up to progression, an average of 1 year
  The time interval between study entry and date of progression (using RECIST 1.1)
Overall survival | Through study completion, an average of 12 months
  The time interval between study entry and death from any cause
Tumor response | Immediately after each cycle of treatment, up to progression, an average of 1 year
  Using CT-scan or MRI imaging (using RECIST 1.1)
Adverse events | Through study completion, an average of 12 months (plus 30 days)
  The adverse events (AE) are collected to evaluate the safety of the study treatment.
The feasibility of evaluated therapy | Through study completion, an average of 12 months
  assessed in terms of frequency of dose reductions or temporary stops of treatment
Quality of life of the patient (KindL) | Baseline, week 7 and week 13
  Ravens-Sieberer and Bullinger Quality of Life Questionnaire will be used to measure the quality of life of the patients. The score can go from 0 to 100, and the higher score corresponds to a higher health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Hélène SUDOUR-BONNANGE, MD, Principal Investigator — Centre Oscar Lambret; Arnauld VERSCHUUR, MD, PhD, Principal Investigator — CHU La Timone
Locations (18):
- France (18):
  - CHU Amiens Picardie, Amiens
  - CHU de Besancon, Besançon
  - CHRU de Bordeaux Hôpital des Enfants, Bordeaux
  - CHU GRENOBLE ALPES - Hôpital COUPLE ENFANT, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital pour Enfants " La Timone " AP-HM, Marseille
  - CHU de MONTPELLIER - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU Nantes, Nantes
  - CHU de Nice - Hôpital Archet 2, Nice
  - Hôpital Armand-TROUSSEAU, Paris
  - CHU Hôpital Sud, Rennes
  - Chu Rouen, Rouen
  - CHU La Réunion, Saint-Denis
  - CHRU Strasbourg - Hôpital de Hautepierre, Strasbourg
  - CHU Toulouse - Hôpital des Enfants, Toulouse
  - CHRU NANCY - Hôpital d'Enfants, Vandœuvre-lès-Nancy
  - Gustave ROUSSY, Villejuif

IPD SHARING:
Plan to Share IPD: No